CLINICAL TRIAL: NCT01515215
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Treatment Resistant Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 040 / 2008
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depression Disorder; Treatment Resistance; repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-frequency Left rTMS (Active Comparator): Intensity: rTMS treatment intensity determined by using resting motor threshold (RMT). Treatment will be delivered at 120% of the RMT.
  Site of Stimulation: left hemisphere of DLPFC.
  Frequency: 10 Hz.
  Duration: 42 Trains, 5 second duration, 25 second inter-train interval.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Bilateral rTMS (Active Comparator): Intensity: rTMS treatment intensity determined by the RMT. Treatment will be delivered at 120% of the RMT.
  Sites of Stimulation: right and left hemispheres of the DLPFC.
  Frequency: 1 Hz over the right DLPFC followed by 10 Hz over the left DLPFC.
  Duration: right: 1 Train of 600 pulses; left: 30 Trains, 5 second duration, 25 second inter-train interval.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham rTMS Treatment is applied as either Bilateral rTMS or HFL-rTMS (randomly assigned), but with the coil angled 90 degrees away from the skull in a single-wing tilt position. This method produces sound and some somatic sensation (e.g., contraction of scalp muscles) similar to those of active stimulation, but with minimal direct brain effects.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Magnetic pulses to specific brain regions. (MagPro X100)
  Other Names: MagPro X100 Series (Magventure A/S, Farum, Denmark)

SUMMARY:
Major Depressive Disorder (MDD) is one of the most prevalent mental illnesses in North America, in which 30% - 40% fail to respond to conventional treatment. Repetitive Transcranial Magnetic Stimulation (rTMS) has been shown to be an effective therapeutic tool for the treatment of MDD. This form of treatment involves a series of magnetic pulses directed to the brain for about 30 minutes. Importantly, such treatment is very safe and well tolerated. However, to date, most treatment studies show modest efficacy due to limitations, including: 1) treatments that are delivered to only one side of the brain; 2) treatment that does not directly target a specific brain region associated with depression; 3) treatments that are of short duration; 4) treatments that are of insufficient intensity; and 5) insufficient understanding of the brain mechanisms responsible for therapeutic effect. This study is designed to directly address all of these limitations, as well as explore brain mechanisms (e.g. cortical excitability) through which treatment is optimized.

DETAILED DESCRIPTION:
Several studies have demonstrated that rTMS is an efficacious treatment for treatment resistant major depressive disorder (TRD). However, recent meta-analyses, and more recent, large, multi-centre studies, have provided evidence suggesting that rTMS, at best, provides modest therapeutic efficacy compared to sham stimulation.

Several reasons may account for this modest therapeutic effect. First, the majority of these studies involved left-sided treatment alone to the dorsolateral prefrontal cortex (DLPFC), which is a significant limitation when considering that electroconvulsive therapy - another form of brain stimulation used in TRD - has been shown to be less efficacious when used unilaterally, compared to bilaterally.

Second, sub-optimal methods were utilized to target the DLPFC (i.e., '5-cm anterior method'), limiting the treatment potential of what is inherently a targeted form of treatment. In this regard, recent data from the investigators suggests that treatment directly targeting the DLPFC provides enhanced therapeutic efficacy compared to the '5-cm anterior' method.

Third, treatment durations were typically short (i.e., 2-4 weeks). Fourth, stimulation intensity may have been insufficient by not taking into consideration coil-to-cortex distance, which is of particular importance when considering that this parameter may contribute significantly to rTMS-induced antidepressant response. Fifth, there has not been a study that has examined TRD across the lifespan in a way that addresses the differences between older and younger adults. Therefore, the investigators propose to conduct a study evaluating the efficacy of rTMS for TRD that directly addresses all 5 of these major limitations.

This study will compare bilateral rTMS to unilateral rTMS and will involve targeting the DLPFC using cortical co-registration techniques, as well as treatments of optimal duration (i.e., up to 6 weeks) and intensity parameters (i.e., adjusted for coil-to-cortex distance). The use of distance cortical co-registration and adjustment for coil-to-cortex distance addresses the major limitation (lack of stimulation intensity to compensate for age-related prefrontal atrophy) in studies that have examined rTMS in an elderly sample. Preliminary data from this research group provide compelling evidence that rTMS may, indeed, be effective when some of these limitations are optimized in both younger and older adults. Finally, it is also essential that research investigate the mechanisms of therapeutic efficacy, so that increases in understanding can be translated into enhanced treatment. For several reasons, cortical excitability may represent a neurophysiological process through which the therapeutic effects of rTMS are mediated. Recent advances in electroencephalography (EEG) technology now permit direct measurement of excitability from the DLPFC; thus, we are now able to ascertain whether these are mechanisms through which the therapeutic effects of rTMS in TRD are mediated.

Hypotheses:

Hypothesis 1: Treatment with bilateral and high frequency left rTMS (HFL-rTMS) will both result in a greater reduction in 17-item Hamilton Depression Rating Scale (HAM-D17) scores compared to sham rTMS.

Hypothesis 2: Bilateral rTMS will result in a significantly greater number of patients reaching criteria for therapeutic response and remission on the HAM-D17 compared to unilateral or sham rTMS.

Hypothesis 3: An increase of excitability following HFL-rTMS to the left DLPFC (in the case of bilateral rTMS or HFL-rTMS) and a decrease in excitability following low frequency right-rTMS (LFR-rTMS; in the case of bilateral rTMS) to the right DLPFC will mediate the relationship between rTMS and response in TRD. Finally, the induction of gamma activity following rTMS will be associated with improved treatment efficacy.

Hypothesis 4: rTMS will result in improved executive function in patients over age 60 with TRD.

ELIGIBILITY:
Inclusion Criteria:

* voluntary and competent to consent
* diagnosis of MDD, as confirmed by the Structured Clinical Interview for the DSM-IV (SCID-IV)
* 18 - 85 years of age
* failed to achieve clinical response, or did not tolerate, at least 2 separate antidepressant trials of sufficient dosage for at least 6 wks
* have a score of 20 or greater on the HAM-D17
* have not had an increase or initiation of any psychoactive therapy in the 4 wks prior to testing
* if a woman of childbearing potential, must be on an effective means of birth control

Exclusion Criteria:

* history of DSM-IV confirmed diagnosis of substance dependence in the last 6 months, or substance abuse in the last month
* concomitant, major, unstable medical or neurologic illness
* history of seizures
* acutely suicidal and/or homicidal
* pregnant
* have metal implants
* history of psychosurgery
* co-morbid diagnosis of borderline and/or antisocial personality disorder. as confirmed by the SCID for Axis II Disorders (SCID-II)
* are currently (or in the past 4 weeks) taking more than 2 mg of lorazepam, or equivalent, daily
* ECT treatment in the current episode

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Degree of Change in HAM-D17 Scores | At weeks 3 and/or 6

SECONDARY OUTCOMES:
Degree of Change in Montgomery-Asberg Depression Rating Scale Scores | At weeks 3 and/or 6
Degree of Change in Beck Depression Inventory Scores | At weeks 3 and/or 6
Degree of Change in Brief Psychiatric Ratings Scale Scores | At weeks 3 and/or 6
Changes in Cortical Excitability | At weeks 3 and/or 6
  Assessed via TMS-EEG protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Z. Jeffrey Daskalakis, MD, PhD., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hadas I, Sun Y, Lioumis P, Zomorrodi R, Jones B, Voineskos D, Downar J, Fitzgerald PB, Blumberger DM, Daskalakis ZJ. Association of Repetitive Transcranial Magnetic Stimulation Treatment With Subgenual Cingulate Hyperactivity in Patients With Major Depressive Disorder: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2019 Jun 5;2(6):e195578. doi: 10.1001/jamanetworkopen.2019.5578. PMID 31167023
- [Derived] Trevizol AP, Goldberger KW, Mulsant BH, Rajji TK, Downar J, Daskalakis ZJ, Blumberger DM. Unilateral and bilateral repetitive transcranial magnetic stimulation for treatment-resistant late-life depression. Int J Geriatr Psychiatry. 2019 Jun;34(6):822-827. doi: 10.1002/gps.5091. Epub 2019 Apr 8. PMID 30854751
- [Derived] Voineskos D, Blumberger DM, Zomorrodi R, Rogasch NC, Farzan F, Foussias G, Rajji TK, Daskalakis ZJ. Altered Transcranial Magnetic Stimulation-Electroencephalographic Markers of Inhibition and Excitation in the Dorsolateral Prefrontal Cortex in Major Depressive Disorder. Biol Psychiatry. 2019 Mar 15;85(6):477-486. doi: 10.1016/j.biopsych.2018.09.032. Epub 2018 Oct 18. PMID 30503506
- [Derived] Weissman CR, Blumberger DM, Brown PE, Isserles M, Rajji TK, Downar J, Mulsant BH, Fitzgerald PB, Daskalakis ZJ. Bilateral Repetitive Transcranial Magnetic Stimulation Decreases Suicidal Ideation in Depression. J Clin Psychiatry. 2018 May/Jun;79(3):17m11692. doi: 10.4088/JCP.17m11692. PMID 29701939
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research